CLINICAL TRIAL: NCT00006134
Title: Study of the Predictors of the Course and Early Outcome of Patients With Systemic Lupus Erythematosus: Nature Versus Nurture
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Alabama at Birmingham (Other)
Other Study IDs: 199/15328; UAB-GCRC-617
Record Dates: First submitted 2000-08-03; First posted 2000-08-04 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: arthritis & connective tissue diseases; immunologic disorders and infectious disorders; rare disease; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis; Connective Tissue Diseases; Immune System Diseases; Communicable Diseases; Rare Diseases

SUMMARY:
OBJECTIVES: I. Continue yearly ascertainment visits of all patients of the established Lupus in Minority Populations: Nature vs Nurture (LUMINA) study cohort.

II. Recruit into the LUMINA cohort newly diagnosed patients with systemic lupus erythematosus (SLE).

III. Determine the impact of additional major histocompatibility complex (MHC) and non-MHC genetic factors not previously examined, specifically tumor necrosis factor, mannose binding protein, interleukin-1 receptor antagonist, and bcl-2, on the course and outcome of SLE.

IV. Refine the assessment of those clinical and behavioral-cultural factors found to be important predictors of disease activity, damage, and functioning, thus far in these patients.

V. Determine the relationships among disease activity, disease damage, and physical and mental functioning in these patients as the SLE progresses and the factors that predict them.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a parallel, follow up study of a natural history study. Patients are stratified according to ethnicity (Caucasian vs African-American vs Hispanic).

Patients are examined at baseline and then every 6 months thereafter in order to determine the relative impact of genetic, sociodemographic, and behavioral-cultural factors on disease outcome. Patients are assessed for the following outcome variables: disease activity by the Systemic Lupus Activity Measure (SLAM), disease damage by the Systemic Lupus International Collaborative Clinics Damage Index (SDI), and physical and mental functioning by the Medical Outcomes Study 36 Item Short-Form Health Survey (SF-36). Patients are also assessed for independent variables belonging to the following domains: socioeconomic-demographic, clinical, immunogenetic, and behavioral-cultural. Patients undergo genetic analysis utilizing polymerase chain reaction and electrophoresis to further study the immunogenetic domain and genetic markers that may be related to disease. Specifically, patients' blood is analyzed for tumor necrosis factor alpha, tumor necrosis factor beta, mannose binding protein, interleukin-1 receptor antagonist, and bcl-2.

ELIGIBILITY:
* All systemic lupus erythematosus (SLE) patients currently constituting the established Lupus in Minority Populations: Nature vs Nurture (LUMINA) cohort OR New recruits meeting at least 4 of the 1997 American College of Rheumatology criteria for the classification of SLE
* Disease onset within the past 5 years
* African-American, Hispanic, or Caucasian Self stated, plus the same for all 4 grandparents
* No concurrent participation in any intervention studies
* Not pregnant
* Not mentally retarded
* No prisoners
* No other concurrent disability that would preclude study

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 1993-09

CONTACTS AND LOCATIONS:
Overall Officials: Graciela S. Alarcon, Study Chair — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas Health Science Center - Houston, Houston, Texas